CLINICAL TRIAL: NCT02452333
Title: Oncoplastic Approach to Excisional Breast Biopsies: A Prospective Randomized Controlled Trial
Brief Title: Oncoplastic Approach to Excisional Breast Biopsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 70904504
Record Dates: First submitted 2015-05-18; First posted 2015-05-22 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Neoplasm of Female Breast; Breast Neoplasms Diagnosis; Breast Diseases; Deformity of Reconstructed Breast
Keywords: Excisional breast biopsy; Oncoplastic surgery; Oncoplastic reconstruction; Breast conserving surgery; Tezel method of breast volume measurement
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Evidence-based Oncoplastic Algorithm (Experimental): Oncoplastic Approach Excisional Breast Biopsy, Tezel Method of Breast Volume Measurement and Cosmetic Assessment
  Interventions: Procedure: Oncoplastic Approach Excisional Breast Biopsy; Other: Tezel Method of Breast Volume Measurement; Other: Cosmetic Assessment
- Control (Experimental): - Conventional Excisional Breast Biopsy, Tezel Method of Breast Volume Measurement and Cosmetic Assessment
  Interventions: Procedure: Conventional Excisional Breast Biopsy; Other: Tezel Method of Breast Volume Measurement; Other: Cosmetic Assessment

INTERVENTIONS:
Procedure: Oncoplastic Approach Excisional Breast Biopsy — Evidence based quadrant by quadrant oncoplastic algorithm reinforced with videoscopic applications for peripheral lesions.
  Arms: Evidence-based Oncoplastic Algorithm
Procedure: Conventional Excisional Breast Biopsy — Conventional Excisional Breast Biopsy
  Arms: Control
Other: Tezel Method of Breast Volume Measurement — Tezel Method is a simple, accurate and non-invasive method of measuring differences in breast volume based on Archimedes' principle
Other: Cosmetic Assessment — Cosmetic Assessment with Harris scale graded by patient, surgeon and professional third party. A standardised photograph of front, side and mediolateral oblique views will be taken using a digital camera for professional third party observers.

SUMMARY:
Many studies focusing on breast conserving surgery have affirmed the cosmetic effectiveness and oncologic success of oncoplastic methods and even modified variants of these methods reinforced with videoscopic applications. However, primary lumpectomy subjects in these studies are mainly patients who have already received the diagnosis of malignancy before the surgery. There is not much comprehensive work reported for patients without the diagnosis of malignancy. In this regard, the investigators believe the intent of the innovative oncoplastic intervention to the breast is underestimated in terms of providing diagnosis simultaneously constituting the basic component of surgical treatment. Thus, the purpose of this prospectively planned study is to provide and investigate the outcomes of an evidence-based oncoplastic approach algorithm for excisional breast biopsies.

DETAILED DESCRIPTION:
Excisional breast biopsy is one of the routine surgical interventions in general surgery clinics, implemented for clinical diagnosis of suspicious breast lesions. It is the diagnostic method of choice especially when fine needle aspiration biopsy (FNA), core cutting needle (trucut) biopsy or vacuum-assisted core biopsy as part of a non-invasive approach can not provide sufficient diagnostic efficiency for the diagnosis of non-palpable breast lesions. This invasive biopsy approach must be selectively tailored according to the nature of the lesion, either directly or as a second-stage procedure, necessarily, if a sufficiently precise diagnosis cannot be reached after practicing less-invasive protocols. By definition, basic difference from a segmental mastectomy or a lumpectomy is that excisional breast biopsy is a surgical procedure to remove suspicious breast tissue and a small amount of normal tissue around it only before the pathologic diagnosis is confirmed.

Prebiopsy localisation modalities like wire-guidance or radioisotope occult lesion localization (ROLL) are proven to reduce the rates of margin positivity at initial lumpectomies in breast cancer. Accomplishing the excision as a whole with a 1 cm layer of normal tissue around by means of an incision confined to possible mastectomy line, whilst preserving the skin if it is 1cm far away from the suspicious area and a three-dimensional marking on the specimen are considered to be general principles in conventional excisional breast biopsies. In the same way, another ground rule would be close collaboration with plastic and reconstructive surgery department, especially when significant relative breast volume loss is anticipated and defect should be restored using volume replacement methods or when the nipple and areola complex (NAC) is under threat. It is imperative that the patient be informed of the common risks and reasonable alternatives to the proposed treatment. For patients seeking additional advice on NAC disturbances it is important to keep in mind that the tattoo art might be an appealing suggestion; many consider tattooing as a practical complementary solution for sequela after reconstruction of Nipple-areolar complex.

On the other hand, in the vast majority of the cases the mainstay of treatment does not entail surgical resection of NAC or requisite volume replacement, but still there is debate as to whether surgeons should place parenchymal sutures to approximate the cut edges of the cavity walls. The rationale behind this debate is that closure of the tissue defect with direct suture approximation brings about a considerable heterogeneity when it comes to cosmetic parameters. Besides, in many cases, when not coupled with overlying skin dissection after probable dimples observed on the skin while knotting each suture, this modality is ended up too far off target to merit the highest degree of patient satisfaction. Fortunately, surgical algorithms for breast tumors have been refined a great deal in recent years with rapid developments and key technique definitions in the field of oncoplastic surgery and opinions favoring parenchymal sutures have been strengthened.

Many studies focusing on breast conserving surgery have affirmed the cosmetic effectiveness and oncologic success of oncoplastic methods and even modified variants of these methods reinforced with videoscopic applications. However, primary lumpectomy subjects in these studies are mainly patients who have already received the diagnosis of malignancy before the surgery. There is not much comprehensive work reported for patients without the diagnosis of malignancy. In this regard, the investigators believe the intent of the innovative oncoplastic intervention to the breast is underestimated in terms of providing diagnosis simultaneously constituting the basic component of surgical treatment. Thus, the purpose of this prospectively planned study is to provide and investigate the outcomes of an evidence-based oncoplastic approach algorithm for excisional breast biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are decided to be suitable for excisional breast biopsy.
* Nonpalpable breast lesions suspicious for malignancy where less-invasive approach like fine needle aspiration biopsy (FNA), core cutting needle (trucut) biopsy or vacuum-assisted core biopsy can not provide sufficient diagnostic efficiency for the diagnosis.
* Palpable breast lesions when a sufficiently precise diagnosis cannot be reached after practicing less-invasive protocols.

Exclusion Criteria:

* Patients who are decided to be suitable for mastectomy included protocols as the primary surgery.
* Patients who have previously had breast surgery.
* Patients who refused excisional breast biopsy.
* Patients who do not want to be photographed for cosmetic evaluations.
* Patients diagnosed with secondary suspicious breast lesions necessitating surgical intervention during the follow-up period.
* Presence of probable multicentric lesions.
* Refusal of the patient to participate in the study for any reason.
* Aberrations in the normal development and involution of the breast
* Injury or trauma history of the breast resulted in deformity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Harris scale for the cosmetic result. | 3 months
  Patient, surgeon and professional third party observers rate cosmetic results (in terms of color, symmetry, contour and general cosmetic outcome) on a four-point scale:
  (4) excellent-treated breast nearly identical to untreated breast; (3) good-treated breast slightly different from untreated; (2) fair-treated breast clearly different from untreated but not seriously distorted; (1) poor- treated breast seriously distorted.

SECONDARY OUTCOMES:
Surgical margin positivity for malignancy | Approximately 2 weeks
  Ultimate histopathologic diagnosis
Radiologic assessment of surgical margins | Intraoperatively assessed
  Specimen mammography: Applicable to mammographically depicted lesions only
Morbidity | 3 months
  Bleeding, hematoma, seroma, necrosis or infection after surgery.
Reoperations | 3 months
  Need for any reoperations whether morbidity or surgical margins related.
Breast Size | Preoperatively assessed
  Unilateral breast volume measured with Tezel method to discriminate small (250 cc and less) vs. medium/large (>250 cc) breasts; determine oncoplastic intervention level (I or II) after assessment of anticipated volume ratio of the resection specimen.
Lesion Peripherality | Preoperatively assessed
  Lesion peripherality along with the videoscopic application preference is decided after assessment of areolar diameter, distance between areolar margin and the skin projection of the central spot of the lesion together with the depth of the lesion; all of which are determinants for ease of access to resection area.
Anticipated specimen volume | Preoperatively assessed
  Preoperatively anticipated specimen volume according to radiologic investigation.
Exact specimen volume | Intraoperatively assessed
  True volume of the excised breast tissue

CONTACTS AND LOCATIONS:
Overall Officials: Cumhur Arıcı, Professor, Study Director — Akdeniz University, General Surgery Department
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Santos G, Urban C, Edelweiss MI, Zucca-Matthes G, de Oliveira VM, Arana GH, Iera M, Rietjens M, de Lima RS, Spautz C, Kuroda F, Anselmi K, Capp E. Long-Term Comparison of Aesthetical Outcomes After Oncoplastic Surgery and Lumpectomy in Breast Cancer Patients. Ann Surg Oncol. 2015 Aug;22(8):2500-8. doi: 10.1245/s10434-014-4301-6. Epub 2014 Dec 18. PMID 25519931
- [Background] McCulley SJ, Macmillan RD. Planning and use of therapeutic mammoplasty--Nottingham approach. Br J Plast Surg. 2005 Oct;58(7):889-901. doi: 10.1016/j.bjps.2005.03.008. PMID 16043150
- [Background] Clough KB, Ihrai T, Oden S, Kaufman G, Massey E, Nos C. Oncoplastic surgery for breast cancer based on tumour location and a quadrant-per-quadrant atlas. Br J Surg. 2012 Oct;99(10):1389-95. doi: 10.1002/bjs.8877. PMID 22961518
- [Background] Cardoso MJ, Cardoso JS, Wild T, Krois W, Fitzal F. Comparing two objective methods for the aesthetic evaluation of breast cancer conservative treatment. Breast Cancer Res Treat. 2009 Jul;116(1):149-52. doi: 10.1007/s10549-008-0173-4. Epub 2008 Sep 7. PMID 18777134
- [Background] Yamashita K, Shimizu K. Transaxillary retromammary route approach of video-assisted breast surgery enables the inner-side breast cancer to be resected for breast conserving surgery. Am J Surg. 2008 Oct;196(4):578-81. doi: 10.1016/j.amjsurg.2008.06.028. PMID 18809067
- [Background] Serra-Renom JM, Serra-Mestre JM, Martinez L, D'Andrea F. Endoscopic reconstruction of partial mastectomy defects using latissimus dorsi muscle flap without causing scars on the back. Aesthetic Plast Surg. 2013 Oct;37(5):941-9. doi: 10.1007/s00266-013-0192-3. Epub 2013 Jul 23. PMID 23877754
- [Background] Tezel E, Numanoglu A. Practical do-it-yourself device for accurate volume measurement of breast. Plast Reconstr Surg. 2000 Mar;105(3):1019-23. doi: 10.1097/00006534-200003000-00028. PMID 10724264
- [Background] Nakajima H, Fujiwara I, Mizuta N, Sakaguchi K, Hachimine Y, Magae J. Video-assisted skin-sparing breast-conserving surgery for breast cancer and immediate reconstruction with autologous tissue: clinical outcomes. Ann Surg Oncol. 2009 Jul;16(7):1982-9. doi: 10.1245/s10434-009-0429-1. Epub 2009 Apr 24. PMID 19390899
- [Background] Nakajima H, Fujiwara I, Mizuta N, Sakaguchi K, Hachimine Y. Video-assisted skin-sparing breast-conserving surgery for breast cancer and immediate reconstruction with autologous tissue. Ann Surg. 2009 Jan;249(1):91-6. doi: 10.1097/SLA.0b013e31818e3fa6. PMID 19106682
- [Background] Zaha H. Partial breast reconstruction for the medial quadrants using the omental flap. Ann Surg Oncol. 2014 Oct;21(10):3358. doi: 10.1245/s10434-014-3907-z. Epub 2014 Jul 26. PMID 25063006
- See also: Oncoplastic approach to excisional breast biopsies: a randomized controlled, phase 2a trial — https://dx.doi.org/10.1007/s12282-018-0892-2